CLINICAL TRIAL: NCT03743272
Title: Repeatability and Reproducibility of Multiparametric MRI (LiverMultiScan)
Brief Title: Repeatability and Reproducibility of Multiparametric MRI
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: LMSRR
Record Dates: First submitted 2018-11-08; First posted 2018-11-16 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Liver Diseases; Primary Biliary Cirrhosis; Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis; Cirrhosis; Hemochromatosis; Viral Hepatitis; Autoimmune Hepatitis; Primary Sclerosing Cholangitis
Keywords: Multiparametric MRI; LiverMultiScan; Repeatability; Reproducibility; Liver MRI
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis, Biliary; Non-alcoholic Fatty Liver Disease; Fibrosis; Hemochromatosis; Hepatitis, Autoimmune; Cholangitis, Sclerosing | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Liver condition: Participants who have a history of of liver disease
  Interventions: Device: LiverMultiScan
- Healthy volunteers: Participants who have do not have a diagnosed liver condition and are in general good health
  Interventions: Device: LiverMultiScan

INTERVENTIONS:
Device: LiverMultiScan — Up to 6 separate 5-10 minute abdominal MRI scans. Each scan requires a short breath hold.
  Other Names: Multiparametric Magnetic Resonance Imaging (mpMRI)

SUMMARY:
This study aims to prospectively assess the repeatability and reproducibility of iron-corrected T1 (cT1), T2*, and hepatic proton density fat fraction (PDFF) quantification with multiparametric MRI using the LiverMultiScan™ (LMS, Perspectum Diagnostics, Oxford, UK) protocol across different field strengths, scanner manufacturers and models.

DETAILED DESCRIPTION:
As the burden of liver disease reaches epidemic levels, there is a high unmet medical need to develop robust, accurate and reproducible non-invasive methods to quantify liver tissue characteristics for use in clinical development and ultimately in clinical practice. Repeatability and reproducibility validation studies are important in evaluating metrics, such that any changes can be confidently attributed to disease progression or regression, rather than inter-examination variability in the instrument.

Magnetic resonance (MR) techniques offer an attractive non-invasive option for liver assessment. Multiparametric MRI is a safe and non-invasive method for quantification of liver tissue characteristics. Images for quantification of hepatic fat from proton density fat fraction (PDFF) maps, T2*, and iron-corrected T1 (cT1) can be rapidly obtained during abdominal breath-hold acquisitions without the need for contrast agents or additional external hardware. Iron correction of T1 is necessary to address the confounding effects of excess iron, which is common in chronic liver disease. LiverMultiScan™ (LMS, Perspectum Diagnostics, Oxford, UK) is a software application that can be used with supported MR-systems to correct T1 for the effects of excess iron, and thus, to calculate cT1 from T1 and T2* maps, and standardise to a 3T field strength.

This method has been shown to have high diagnostic accuracy for the assessment of liver fibrosis compared to histology, predict clinical outcomes in patients with mixed liver disease aetiology, stratify patients with non-alcoholic steatohepatitis (NASH) and cirrhosis, reliably exclude clinically significant liver disease and is cost-effective in diagnosing NAFLD.

In addition to demonstrating accuracy, imaging biomarker validation requires precision and repeatability (US Department of Health and Human Services, 2015). From a clinical perspective, it is essential to ensure that there is good inter-examination repeatability, so that any changes seen can be correctly attributed to disease progression or regression, rather than inter-examination variability. This is tested by examining the closeness of repeated measurements made in different MR examinations (with both subject and coil repositioning) over a time frame in which physiologic conditions are assumed constant.

This study aims to systematically test the repeatability and reproducibility of each multiparametric MRI measurement, cT1, T2* and PDFF, corresponding to hepatic fibro-inflammation, iron and fat respectively, across scanner field strength, manufacturer and model in human participants and phantoms.

ELIGIBILITY:
Inclusion Criteria:

* Any person over 18 years of age.
* Participant is willing and able to give informed consent.

Exclusion Criteria:

* The participant may not enter the study if they have any contraindication to magnetic resonance imaging (inc pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study or affect the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are those with mixed liver disease aetiology and those without any history of liver disease in order to represent a wide range of values of hepatic fat, iron, and fibro-inflammatory status.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-06-03 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Repeatability | 2 years
  Comparison of multi-parametric MRI measures (MRI-PDFF, T2* and iron-corrected T1 (cT1)) from repeated acquisitions of the same participant on the same scanner.
Reproducibility | 2 years
  Comparison of multi-parametric MRI measures (MRI-PDFF, T2* and iron-corrected T1 (cT1)) from repeated acquisitions of the same participant on different scanners (1.5T and 3.0T).

CONTACTS AND LOCATIONS:
Overall Officials: Rajarshi Banerjee, BM BCh MS DPhil, Principal Investigator — Perspectum Diagnostics
Locations (4):
- Leiden University Medical Centre, Leiden, Netherlands
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - University of Oxford Centre for Clinical Magnetic Resonance Research (OCMR), Oxford, Oxfordshire
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pickles E, Kumar S, Brady M, Telford A, Pavlides M, Bulte D. Comparison of liver iron concentration calculated from R2* at 1.5 T and 3 T. Abdom Radiol (NY). 2023 Mar;48(3):865-873. doi: 10.1007/s00261-022-03762-4. Epub 2022 Dec 15. PMID 36520162